CLINICAL TRIAL: NCT06108037
Title: Duke Health Listens Survey on Generative Artificial Intelligence (AI) for MyChart Messaging
Brief Title: DHL Survey on Generative AI for MyChart Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00113587
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-10

CONDITIONS: Communication
Keywords: Artificial Intelligence; Generative Artificial Intelligence
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: * Participants will be randomly allocated to one of six arms.
  * Over the course of the study period, there will be multiple rounds of surveys, which will consist of a clinical scenario, a response (human or AI generated), and a disclosure statement (none, human, or AI).
  * All respondents within an arm will be assigned to a sequence of response-disclosure pairs prior to the first round of surveys.
Who Masked: Participant
Masking Description: Participants will not be aware of the arm they are assigned to. There is no care provider or outcomes assessor in this study, as the patients will report their own perceptions in a survey.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A (Other): Each arm will receive 3 clinical scenarios spaced over time across 3 Sends. The 6 groups (Arms A-F) will be arranged with naming conventions as such:
  * First letter = A, B, or C where A = scenario 1, B = scenario 2, and C = scenario 3.
  * Second letter(s) = H or AI, where H = human response and AI = AI-written response to the patient question posed.
  * Third letter(s) = N, C, or H, where N = no disclosure, C = computer disclosure, and H = human disclosure. This refers to the disclosure at the bottom of the response message whereby the author is or is not disclosed.
  Arm A receives AHN in Send 1, BAIC in Send 2, and CHH in Send 3
  Interventions: Behavioral: Generative AI for electronic communication and disclosure
- Arm B (Other): Each arm will receive 3 clinical scenarios spaced over time across 3 Sends. The 6 groups (Arms A-F) will be arranged with naming conventions as such:
  * First letter = A, B, or C where A = scenario 1, B = scenario 2, and C = scenario 3.
  * Second letter(s) = H or AI, where H = human response and AI = AI-written response to the patient question posed.
  * Third letter(s) = N, C, or H, where N = no disclosure, C = computer disclosure, and H = human disclosure. This refers to the disclosure at the bottom of the response message whereby the author is or is not disclosed.
  Arm B receives BHC in Send 1, CAIH in Send 2, and AAIN in Send 3
  Interventions: Behavioral: Generative AI for electronic communication and disclosure
- Arm C (Other): Each arm will receive 3 clinical scenarios spaced over time across 3 Sends. The 6 groups (Arms A-F) will be arranged with naming conventions as such:
  * First letter = A, B, or C where A = scenario 1, B = scenario 2, and C = scenario 3.
  * Second letter(s) = H or AI, where H = human response and AI = AI-written response to the patient question posed.
  * Third letter(s) = N, C, or H, where N = no disclosure, C = computer disclosure, and H = human disclosure. This refers to the disclosure at the bottom of the response message whereby the author is or is not disclosed.
  Arm C receives CHC in Send 1, AHH in Send 2, and BAIN in Send 3
  Interventions: Behavioral: Generative AI for electronic communication and disclosure
- Arm D (Other): Each arm will receive 3 clinical scenarios spaced over time across 3 Sends. The 6 groups (Arms A-F) will be arranged with naming conventions as such:
  * First letter = A, B, or C where A = scenario 1, B = scenario 2, and C = scenario 3.
  * Second letter(s) = H or AI, where H = human response and AI = AI-written response to the patient question posed.
  * Third letter(s) = N, C, or H, where N = no disclosure, C = computer disclosure, and H = human disclosure. This refers to the disclosure at the bottom of the response message whereby the author is or is not disclosed.
  Arm D receives AAIH in Send 1, BHN in Send 2, and CAIC in Send 3
  Interventions: Behavioral: Generative AI for electronic communication and disclosure
- Arm E (Other): Each arm will receive 3 clinical scenarios spaced over time across 3 Sends. The 6 groups (Arms A-F) will be arranged with naming conventions as such:
  * First letter = A, B, or C where A = scenario 1, B = scenario 2, and C = scenario 3.
  * Second letter(s) = H or AI, where H = human response and AI = AI-written response to the patient question posed.
  * Third letter(s) = N, C, or H, where N = no disclosure, C = computer disclosure, and H = human disclosure. This refers to the disclosure at the bottom of the response message whereby the author is or is not disclosed.
  Arm E receives BAIH in Send 1, CHN in Send 2, and AHC in Send 3
  Interventions: Behavioral: Generative AI for electronic communication and disclosure
- Arm F (Other): Each arm will receive 3 clinical scenarios spaced over time across 3 Sends. The 6 groups (Arms A-F) will be arranged with naming conventions as such:
  * First letter = A, B, or C where A = scenario 1, B = scenario 2, and C = scenario 3.
  * Second letter(s) = H or AI, where H = human response and AI = AI-written response to the patient question posed.
  * Third letter(s) = N, C, or H, where N = no disclosure, C = computer disclosure, and H = human disclosure. This refers to the disclosure at the bottom of the response message whereby the author is or is not disclosed.
  Arm F receives CAIN in Send 1, AAIC in Send 2, and BHH in Send 3
  Interventions: Behavioral: Generative AI for electronic communication and disclosure

INTERVENTIONS:
Behavioral: Generative AI for electronic communication and disclosure — We will use a large language model such as GPT 3.5 to automatically generate responses to fictional messages to a physician. We will disclose whether the message was generated using this technology or not. There are 3 clinical scenarios and 6 pairs of human/AI response and human disclosure/AI disclosure/not disclosed that will test patient attitudes toward this technology.

SUMMARY:
The purpose of this study is to understand how patients feel about the use of computer programs to create responses when they send electronic messages to their doctors.

DETAILED DESCRIPTION:
* The investigators will create short surveys online to ask patients how they feel about using computer programs that create messages in their medical records.
* The surveys will show fictional situations where patients ask questions and get answers from either real people or computer programs, with or without a disclosure about how the response was written.
* The investigators will ask the people taking the survey to share what they think about these situations using tools like rating scales, comparison scales, or written responses.
* If patients want to, they can provide their contact information to be part of future discussion groups. Participants do not have to give any personal information to complete the survey.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Duke Health Listens patient advocacy community

Exclusion Criteria:

* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1454 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction, as measured by survey | Up to 2 weeks
  Likert-scale responses to satisfaction question: "I am satisfied with this interaction", on a scale from 1-5 with answer options of Strongly Disagree (1), Disagree (2), Neither agree nor disagree (3), Agree (4), and Strongly agree (5).
Patient attitudes towards utility, as measured by survey | Up to 2 weeks
  Likert-scale responses to utility question: "The information is useful", on a scale from 1-5 with answer options of Strongly Disagree (1), Disagree (2), Neither agree nor disagree (3), Agree (4), and Strongly agree (5).
Patient empathy, as measured by survey | Up to 2 weeks
  Likert-scale responses to empathy question: "I feel cared for during this interaction", on a scale from 1-5 with answer options of Strongly Disagree (1), Disagree (2), Neither agree nor disagree (3), Agree (4), and Strongly agree (5).

CONTACTS AND LOCATIONS:
Overall Officials: Anand Chowdhury, MD, MMCi, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not collect individual patient identifiers, and aggregate data will be reported

REFERENCES:
- [Background] Ayers JW, Poliak A, Dredze M, Leas EC, Zhu Z, Kelley JB, Faix DJ, Goodman AM, Longhurst CA, Hogarth M, Smith DM. Comparing Physician and Artificial Intelligence Chatbot Responses to Patient Questions Posted to a Public Social Media Forum. JAMA Intern Med. 2023 Jun 1;183(6):589-596. doi: 10.1001/jamainternmed.2023.1838. PMID 37115527